CLINICAL TRIAL: NCT02162914
Title: REGORAFENIB AFTER FAILURE OF GEMCITABINE AND PLATINUM-BASED CHEMOTHERAPY FOR LOCALLY ADVANCED (NON RESECTABLE) AND METASTATIC INTRA-HEPATIC OR HILAR CHOLANGIOCARCINOMA: A Randomized Double-blinded Phase II Trial.
Brief Title: Regorafenib Versus Placebo to Treat Cholangiocarcinoma
Acronym: REACHIN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-005626-30
Record Dates: First submitted 2014-05-26; First posted 2014-06-13 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Cholangiocarcinoma
Keywords: Intra-hepatic; Hilar; Locally Advanced; Non Resectable; Metastatic; Regorafenib; Placebo
MeSH Terms: conditions — Cholangiocarcinoma; Neoplasm Metastasis | interventions — regorafenib; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regorafenib/active (Active Comparator): Subjects randomized to be treated with Regorafenib (active product) will receive once a day 160 mg po (four tablets of 40 mg) for 3 weeks of every 4 weeks cycle (3 weeks on and 1 week off). Duration of one cycle is 28 days.
  Interventions: Drug: Regorafenib/active
- Regorafenib/placebo (Placebo Comparator): Subjects randomized to be treated with Regorafenib (placebo) will receive once a day 160 mg po (four tablets of 40 mg) for 3 weeks of every 4 weeks cycle (3 weeks on and 1 week off). Duration of one cycle is 28 days.
  Interventions: Drug: Regorafenib/placebo

INTERVENTIONS:
Drug: Regorafenib/active — Subjects randomized to be treated with Regorafenib/active will receive once a day 160 mg po (four tablets of 40 mg) for 3 weeks of every 4 weeks cycle (3 weeks on and 1 week off) Duration of one cycle is 28 days
  Arms: Regorafenib/active
Drug: Regorafenib/placebo — Subjects randomized to be treated with Regorafenib/placebo will receive once a day 160 mg po (four tablets of 40 mg) for 3 weeks of every 4 weeks cycle (3 weeks on and 1 week off) Duration of one cycle is 28 days
  Arms: Regorafenib/placebo

SUMMARY:
The study is a multicenter randomized (1:1) placebo-controlled, double-blinded phase II trial aiming to demonstrate an improvement of median PFS when treating locally advanced unresectable or metastatic patients suffering from an intra-hepatic or hilum (mass-forming) cholangiocarcinoma with Regorafenib as compared to placebo, and after progression after GEM-CDDP (or GEM-OX), or gemcitabine alone followed or preceded by platinum (CDDP or oxaliplatin)-based chemotherapy.

The principal objective is to investigate Regorafenib efficacy by prospectively evaluating the PFS after the administration of Regorafenib combined with BSC as compared to placebo with BSC. Hypothesis is a 50% improvement in median PFS (from 6 weeks to 12 weeks in Regorafenib group).

DETAILED DESCRIPTION:
The principal objective is to investigate Regorafenib efficacy by prospectively evaluating the PFS after the administration of Regorafenib combined with BSC as compared to placebo with BSC. Hypothesis is a 50% improvement in median PFS (from 6 weeks to 12 weeks in Regorafenib group).

ELIGIBILITY:
Inclusion Criteria:

* histologically proven intra-hepatic or hilum cholangiocarcinoma (mass forming, not "liniting" tumor), locally advanced unresectable or metastatic
* progression documented after GEM-CDDP (or GEM-OX), or gemcitabine alone followed or preceded by platinum-based (CDDP or oxaliplatin) chemotherapy
* age > 18 years
* ECOG PS 0/1 at study entry
* measurable disease according to RECIST version 1.1
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirementsconducted within 7 days of starting to study treatment:

oSerum creatinine <1.5x upper reference range

oTotal bilirubin <1.5x ULN

oAlanine transaminase (ALT) and aspartate aminotransferase (AST) < 2.5x ULN (<5x ULN forpatients with liver involvement of their cancer).

oAmylase and lipase <1.5x ULN.

* life expectancy of at least 12 weeks
* effective contraception for both male and female patients if the risk of conception exists
* negative proteinuria on dipstick or 24 hours proteinuria<1000mg
* signed written informed consent

Exclusion Criteria:

* unability to take oral medication
* any malabsorption condition
* patients taking strong cytochrome P (CYP) CYP3A4 inhibitors (eg. Clarithromycin, indinavir,itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telithromycin,voriconazole) or strong CYP3A4 inducers (eg. Carbamazepine, phenobarbital, phenytoin, rifampin, St-John's Wort) (see section 8)
* persistent proteinuria >3.5g/24 hours measured by urine protein-creatinine ratio from a random urinesample (persistent proteinuria >3 non-healing woud, ulcer, or bone fracture
* any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of studymedication
* interstitial lund disease with ongoing signs and symptoms at the time of informed consent
* uncontrolled concurrent CNS, cardiac, infectious diseases, hypertension
* history of myocardial infarction, deep venous or arterial thrombosis, cerebrovascular accident (CVA) during the last 6 months
* previous exposure to anti-VEGF targeting therapy (including Regorafenib) and to signal transduction inhibitors
* known hypersensitivity to any of the components of study treatments
* previous malignancy in the last past 5 years except basal cell cancer of the skin or preinvasive cancer of the cervix
* pregnant or lactating women, or patients of both genders with procreative potential not using adequate contraceptive methods
* medical or psychological conditions that would not permit the patient to complete the study or sign inform consent
* unstable angina, congestive heart failure ≥NYHA class II
* uncontrolled hypertension despite optimal management (systolic blood pressure >150 mmHg or diastolic pressure > 90mmHg)
* pheochromocytoma
* HIV infection
* active chronic hepatitis B or C with a need for antiviral treatment
* liver failure, cirrhosis Chil Pugh B or C
* brain metastasis
* major surgery, open biopsy or significant traumatic injury within 4 weeks prior to the first dose of treatment
* intra-hepatic locoregional therapy (DC Beads, SIRT)
* history of organ allograft
* ongoing infection
* renal failure requiring dialysis
* patients receiving or having received any investigational treatment within 4 weeks prior to study entry, or participating to another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-03-14 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Improve median PFS | 6 to 12 weeks
  The primary endpoint is to improve median PFS from 6 weeks to 12 weeks in Regorafenib group.

SECONDARY OUTCOMES:
Evaluation of response rate | At pretreatment visit (14 to 1 days before treatment initiation), every 6 weeks for 3 times then every 8 weeks until progression
  -Evaluation of tumor response will be done based on radiological RECIST criteria version 1.1 evaluation (thoraco-abdominal CT scan);
Correlation between radiological response and metabolic response | At pretreatment visit (14 to 1 days before treatment initiation)
  Correlation between radiological response (using RECIST criteria version 1.1) and metabolic response using PET imaging (SUV max modifications). This will only be done if SUV max of the tumor inside the liver at pre-treatment visit is ≥ 175% of the SUV max of the normal liver.
Correlation between radiologic response rate and "Dynamic tumor response rate" | At day 1 (pre-treatment) and day 15 of cycle 1
  Correlation between radiologic response rate (RECIST criteria version 1.1) and "Dynamic tumor response rate". Dynamic response rate is defined by a 20% modification of tumoral perfusion status determined by quantitative DCE-MRI after 14 days of treatment (D1 compared to D15 values);
Correlation between dynamic tumor response rate and metabolic response rate | At cycle 1 day 15
  Correlation between dynamic tumor response rate and metabolic response rate (Pet CT) when first Pet CT is positive
Evaluation of Overall Survival (OS) | After 1 year (March 2015)
  Evaluation of OS at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Demols, MD, PhD, Principal Investigator — Erasme University Hospital
Locations (12):
- Belgium (12):
  - CH Jolimont, Haine-Saint-Paul, Hainaut
  - University Hospitals of Antwerp, Antwerp
  - AZ St-Lucas Brugge, Bruges
  - Erasme University Hospital, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - AZ St-Lucas Gent, Ghent
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - CHC St-Joseph, Liège
  - Hôpital Ambroise Paré, Mons
  - CMSE, Namur

REFERENCES:
- [Derived] Demols A, Borbath I, Van den Eynde M, Houbiers G, Peeters M, Marechal R, Delaunoit T, Goemine JC, Laurent S, Holbrechts S, Paesmans M, Van Laethem JL. Regorafenib after failure of gemcitabine and platinum-based chemotherapy for locally advanced/metastatic biliary tumors: REACHIN, a randomized, double-blind, phase II trial. Ann Oncol. 2020 Sep;31(9):1169-1177. doi: 10.1016/j.annonc.2020.05.018. Epub 2020 May 25. PMID 32464280